CLINICAL TRIAL: NCT01599091
Title: Characterizing Gingival and Periodontal Ligament Fibroblasts Reaction to Infection With the Perio- Pathogenic Bacteria Porphyromonas Gingivalis
Brief Title: Characterizing Gingival and Periodontal Ligament Fibroblasts Reaction to Infection With the Bacteria Porphyromonas Gingivalis
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: GF-PDLF-0148-12-HMO-CTIL; 0148-12-HMO (Other: Hadassah Medical Organization)
Record Dates: First submitted 2012-05-03; First posted 2012-05-15 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2013-09

CONDITIONS: Periodontal Disease
Keywords: Fibroblasts; Periodontal ligament; Gingiva; Porphyromonas gingivalis; Chronic periodontitis; ( patients undergoing tooth extraction will be asked permission to use extracted tooth and gingiva for periodontal disease basic research)
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Anyway extracted teeth and gingiva. Patients undergoing tooth extraction will be asked permission to use the anyway extracted teeth and gingiva in order to harvest fibroblasts for further basic research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fibroblast's donors: Patients undergoing tooth extraction will be asked permission to use the anyway extracted teeth and gingiva in order to harvest fibroblasts for further basic research.
  Interventions: Other: Specimens collection

INTERVENTIONS:
Other: Specimens collection — Tooth extraction will be preformed in the regular way regardless of the study. Patients will be asked permission to obtain the extracted tooth and excess of gingival remnants for further in vitro investigation in the main investigator's laboratory.

SUMMARY:
Porphyromonas gingivalis is one of the major bacteria involved in the formation and progression of chronic periodontitis. Pathogens invading the gingiva face the host's innate immune system at first and later on the acquired immune system which includes secreted antibodies and specialized cells. Although both the arms of the immune system are coordinated to overcome the infection, there are several known mechanisms which help pathogens as Porphyromonas gingivalis evade immunity. As a result, inflammatory mediators secreted by immune cells cause tissue damage and lead the inflammation process towards chronicity instead of clearing the pathogen. Up till recently most of the studies focused on the role of macrophages, dendritic cells and lymphocytes at the response to periodontal pathogenic bacteria while the role of fibroblasts (the most abundant cell in the connective tissue) was less examined. Fibroblasts are spindle shaped cells which have the ability to produce extra cellular matrix and respond to growth factors and cytokines. They are able to affect cells in the infected tissue and contribute to immune response efficiency. As known in the case of lymphocytes, fibroblasts also vary in subtypes, each differs in phenotype, immune interactions, extra cellular matrix production and destruction, migration abilities and so on. Two main fibroblasts subtypes in the oral cavity originate in the gingival tissue and the periodontal ligament anchoring teeth to the surrounding alveolar bone. Amongst the differences between the two are collagen production ability and receptors profile over the cell surface. Considering all that, the investigators aim to obtain and use periodontal ligament and gingival tissues removed anyways during common dental procedures in order to extract the different fibroblasts subtypes residing there and compare their response to Porphyromonas gingivalis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women over 18 years of age, eligible for signing
* Patient in need for a tooth extraction regardless of the study
* Patient understanding and in consent to the character and the purpose of the study
* Patient with healthy gingival and connective tissue surrounding the tooth to be extracted

Exclusion Criteria:

* Pregnant or nursing women. children or non judgemental patients
* Patient undergoing tooth extraction due to periodontitis or any reason related to a problem in the tooth connective tissue
* patient with a Rontgenic bone loss around the tooth to be extracted.
* Patient with any oral disease other than gingivitis.
* Patients with need of pre-medication prior to invasive procedures.
* Patients with background disease or regular use of medications
* Patients treated with antibiotics in the 2 months preceding the tooth extraction.
* Smoking patients.
* Patients with alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healty over 18 years of age eligible for signing patients that go through tooth extraction for reasons not related to the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cytokines, inflammatory mediators and extracellular matrix proteins production and secretion in vitro by fibroblasts | primary outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  healthy patients undergoing tooth extraction will be asked permission to use the anyway extracted tooth and gingiva for basic laboratory research. Periodontal ligament and gingival fibroblasts will be harvested from the collected specimens. Protein production and secretion following in vitro stimulation of the fibroblasts with Porphyromonas gingivalis will be examined to assess their function during periodontal disease.

SECONDARY OUTCOMES:
RNA production in vitro | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  RNA production following in vitro stimulation of fibroblasts with Porphyromonas gingivalis will be examined to assess their function during periodontal disease.
cells motion in vitro | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  fibroblasts and leukocytes (cell line) motion in vitro following co-culture and stimulation with Porphyromonas gingivalis will be examined to assess their function and interactions during periodontal disease
Cytokines, inflammatory mediators and extracellular matrix proteins production and secretion by leukocyte cell lines in vitro | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  fibroblasts and leukocytes (cell line) will be co-cultured with and without Porphyromonas gingivalis stimulation in vitro. Protein production and secretion by leukocytes will be examined to assess their function and interactions with fibroblasts during periodontal disease
RNA production in vitro by leukocyte cell lines | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  fibroblasts and leukocytes (cell line) will be co-cultured with and without Porphyromonas gingivalis stimulation in vitro. RNA production by leukocytes will be examined to assess their function and interactions with fibroblasts during periodontal disease
Bacterial survival | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  Porphyromonas gingivalis survival in vitro following incubation with fibroblasts and leukocytes cell lines (in mono or co-cultures ) will be examined to elucidate cells-bacterial interactions leading to periodontal disease chronicity.
Bacterial adherence to fibroblasts and leukocytes in vitro | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  Porphyromonas gingivalis in vitro adherance to fibroblasts and leukocytes cell lines (in mono or co-cultures ) will be examined to elucidate cells-bacterial interactions leading to periodontal disease chronicity.
cell apoptosis (rate and speed) | outcome will be assessed in vitro within 15 years from specimen collection (basic research)
  in vitro cell apoptosis (rate and speed) will be examined following stimulation with Porphyromonas gingivalis

CONTACTS AND LOCATIONS:
Locations (1):
- : Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Somerman MJ, Archer SY, Imm GR, Foster RA. A comparative study of human periodontal ligament cells and gingival fibroblasts in vitro. J Dent Res. 1988 Jan;67(1):66-70. doi: 10.1177/00220345880670011301. PMID 11039048